CLINICAL TRIAL: NCT02518841
Title: A Comparison of ThermaWedge™ Device and Achilles Tendon Stretching for the Treatment of Plantar Fasciopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jack Taunton, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H14-01870
Record Dates: First submitted 2015-07-13; First posted 2015-08-10 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Plantar Fasciitis; Plantar Fasciopathy
Keywords: ThermaWedge TM; stretches
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Achilles Tendon Stretching (Active Comparator): This is the arm of participants who will first be assigned to perform 6 weeks of achilles tendon stretching as demonstrated in the protocol. As this is a crossover design study, this arm will then switch to 6 weeks of ThermaWedge TM stretching.
  Interventions: Device: ThermaWedge TM; Other: Achilles Tendon Stretching
- ThermaWedge TM (Experimental): This is the arm of participants who will first be assigned to perform 6 weeks of ThermaWedge TM stretching as demonstrated in the protocol. As this is a crossover design study this arm will then switch to 6 weeks of Achilles Tendon Stretching
  Interventions: Device: ThermaWedge TM; Other: Achilles Tendon Stretching

INTERVENTIONS:
Device: ThermaWedge TM — ThermaWedge TM is a foam wedge device that is designed to be used in the treatment of plantar fasciopathy.
Other: Achilles Tendon Stretching — Participants will be asked to perform achilles tendon stretching exercises which will be demonstrated at the initial orientation.

SUMMARY:
The investigators will compare Achilles tendon stretching with a new product called a ThermaWedge™ device, a foam wedge designed to help with certain foot stretches and exercises, in the treatment of chronic plantar fasciopathy. There will be 2 groups each of 25 - 30 participants who have chronic plantar fasciopathy, which is a common cause of foot pain. Exercises will be done for 6 weeks and then each group will do the other exercise protocol for another 6 weeks. Participants will fill out the Foot and Ankle Disability Index scale and numerical analog pain scale and the Global Rating of Change Scale prior to any treatment, weekly during treatment and post treatment. The investigators' hypothesis is that use of the ThermaWedge™ device will result in decreased pain and disability when compared to achilles tendon stretching.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of plantar fasciopathy which has persisted (chronic) for at least 12 months.
* participants need to be able to understand simple instructions about the stretches which will likely include both verbal instructions and pictures and participants need to be able to do all the necessary exercises.
* Participants must have current British Columbia (BC) Medical Service Plan (MSP) health coverage so that if they become injured, they are covered medically.
* Participants must be able to fill out surveys online.
* Participants must also pass a clinical screen where a senior medical student or a physiotherapist, Scott Fraser, will assess the patient for for plantar fasciopathy/fasciitis.

Exclusion Criteria:

* Previous ankle or foot trauma or surgery
* duration of pain of less than 12 months,
* those receiving adjuvant treatment such as injections during the time of the study,
* those who are unable to do the necessary exercises required in the study
* Those who do not have current BC MSP health insurance coverage.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Global Rating of Change Scale - assessing change in pain and function | The participants will use the scale on day 1 of the study, at weeks 1, 2 ,3 ,4 ,5, 6, 7, 8, 9, 10, 11, and 12, as well as 6 and 12 weeks after the completion of the intervention
  This is a rating scale which allows participants to indicate the degree of change in pain/function that the participant has experienced since the start of the intervention
Foot and Ankle Disability Index - assessing change in disability | The participants will use the scale on day 1 of the study, at weeks 1, 2 ,3 ,4 ,5, 6, 7, 8, 9, 10, 11, and 12, as well as 6 and 12 weeks after the completion of the intervention
  This is a questionnaire that assesses the amount of pain and the level of functioning that patient is currently experiencing with respect to the foot and ankle.
Numerical Rating Scale - assessing change in severity of pain | The participants will use the scale on day 1 of the study, at weeks 1, 2 ,3 ,4 ,5, 6, 7, 8, 9, 10, 11, and 12, as well as 6 and 12 weeks after the completion of the intervention
  This is a rating scale on which patients will rate the severity of the worst pain they have experienced in the last week from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taunton, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Digiovanni BF, Nawoczenski DA, Malay DP, Graci PA, Williams TT, Wilding GE, Baumhauer JF. Plantar fascia-specific stretching exercise improves outcomes in patients with chronic plantar fasciitis. A prospective clinical trial with two-year follow-up. J Bone Joint Surg Am. 2006 Aug;88(8):1775-81. doi: 10.2106/JBJS.E.01281. PMID 16882901
- [Background] Ryan M, Hartwell J, Fraser S, Newsham-West R, Taunton J. Comparison of a physiotherapy program versus dexamethasone injections for plantar fasciopathy in prolonged standing workers: a randomized clinical trial. Clin J Sport Med. 2014 May;24(3):211-7. doi: 10.1097/JSM.0000000000000021. PMID 24172656
- [Background] Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID 15134610
- [Background] Ryan M, Fraser S, McDonald K, Taunton J. Examining the degree of pain reduction using a multielement exercise model with a conventional training shoe versus an ultraflexible training shoe for treating plantar fasciitis. Phys Sportsmed. 2009 Dec;37(4):68-74. doi: 10.3810/psm.2009.12.1744. PMID 20048543
- [Background] W. Guy. ECDEU assessment manual for psychopharmacology. Rockville, MD: U.S. Department of Health, Education, and Welfare; 1976.
- [Background] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623